CLINICAL TRIAL: NCT01942681
Title: Multi-institution Study on Efficacy and Safety of Propiverine Hydrochloride for Female Patients With Urge and Stress Urinary Incontinence
Brief Title: Female Patients With Signs of uRgE and Stress Urinary Incontinence Study of Propiverine Hydrochloride
Acronym: FRESH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Shinshu University Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRIGU1309; UMIN000011491 (Other: UMIN Clinical Trials Registry (UMIN-CTR))
Record Dates: First submitted 2013-08-29; First posted 2013-09-16 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Urinary Incontinence
Keywords: female; mixed urinary incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — propiverine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Propiverine Hydrochloride Administration (Other): Administration of Propiverine Hydrochloride for 12 weeks
  Interventions: Drug: Propiverine Hydrochloride

INTERVENTIONS:
Drug: Propiverine Hydrochloride — Administrate Propiverine Hydrochloride for 12 weeks
  Other Names: Bup-4

SUMMARY:
This study is to evaluate the efficacy and safety that the occurrence of incontinence is significantly decrease using the propiverine hydrochloride for 200 female patients with mixed (stress and urge) urinary incontinence in one week during a twelve-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with mixed urinary incontinence (MUI)
2. Patients having symptoms of urinary incontinence for at least 3 months
3. Patients having at least one episode of urge urinary incontinence per week and 4 episodes of stress urinary incontinence per week in a bladder diary.
4. 20 years old or older
5. Patients who meet all the following criteria in ICIQ-SF (1) "2-3 times or more in one week" was selected at Q1. (2) "Small or more" was selected at Q2. (3) "leak at the time of cough or sneeze" or "leak at the time of exercise" was selected at Q4.
6. Less than 100mL of residual urine volume
7. Written informed consent.

Exclusion Criteria:

1. Patients with organ disease such as bladder stones, bladder tumors and urethral stricture in the lower urinary tract
2. Patients with bacterial infections (i.e. bacterial cystitis) or nonbacterial infections (i.e. interstitial cystitis)
3. Patients with advanced lower urinary tract obstruction or urinary retention
4. Patients without urinary sensation
5. Patients with overflow incontinence
6. Patients with history or complications of pelvic organ prolapse
7. Patients with pyloric, duodenal or intestinal obstruction
8. Patients with gastric or intestinal atony
9. Patients with angle-closure glaucoma
10. Patients with myasthenia gravis
11. Patients with severe heart disease
12. Patients with severe constipation
13. Patients with dementia who are not able to complete the questionnaires
14. Patients with history of allergic reaction to Propiverine Hydrochloride or other similar medicine
15. Patients with history of surgery that affect urination such as Trans-Obturator Tape（TOT）or Tension-free Vaginal Tape（TVT）
16. Women who are pregnant, lactating, potentially pregnant or willing to get pregnant
17. Patients with previous surgery of the abdomen and pelvis or radiation within 6 months
18. Patients who started pelvic floor muscle exercise within 3 months
19. Patients who took Propiverine Hydrochloride or other similar medicine within 2 weeks before entry
20. Judged as being unsuitable for the trial by physician.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Occurrence of incontinence | during a twelve-week treatment period
  Change in occurrence of incontinence during a twelve-week treatment

SECONDARY OUTCOMES:
The number of protective pad used | during a twelve-week treatment period
  Change in the number of protective pad used during a twelve-week treatment period
Reduction ratio of the occurrence for incontinence | during a twelve-week treatment period
  Change in reduction ratio of the occurrence for incontinence during a twelve-week treatment period
ICIQ-Short Form(SF) scores | during a twelve-week treatment period
  Change in ICIQ-SF scores during a twelve-week treatment period
I-QOL scores | during a twelve-week treatment period
  Change in I-QOL scores during a twelve-week treatment period
IPSS-QOL scores | during a twelve-week treatment period
  Change in IPSS-QOL scores during a twelve-week treatment period
IPSS symptom scores | during a twelve-week treatment period
  Change in IPSS symptom scores during a twelve-week treatment period
OABSS symptom scores | during a twelve-week treatment period
  Change in OABSS symptom scores during a twelve-week treatment period
Blood pressure | during a twelve-week treatment period
  Change in blood pressure during a twelve-week treatment period
Pulse rate | during a twelve-week treatment period
  Change in pulse rate during a twelve-week treatment period
Safety assessment | during a twelve-week treatment period
  The occurrence of adverse events during a twelve-week treatment period

OTHER OUTCOMES:
Maximum urethral closure pressure | during a twelve-week treatment period
  Change in maximum urethral closure pressure during a twelve-week treatment period
Functional profile length | during a twelve-week treatment period
  Change in functional profile length during a twelve-week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Osamu Nishizawa, M.D., Ph.D., Principal Investigator — Shinshu University Hospital
Locations (1):
- Shinshu University Hospital, Matsumoto, Nagano, Japan